CLINICAL TRIAL: NCT05650788
Title: Exploration of Differences in Metabolite Concentrations by NMR Spectroscopy in the Ventral Striatum, Anterior Cingulate Cortex and Prefrontal Cortex in Euthymic Patients With Unipolar and Bipolar Type II Mood Disorders, as Well as in Healthy Subjects
Acronym: RMN-UNIBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2019 ALLAUZE; 2019-A02607-50 (Other: 2019-A02607-50)
Record Dates: First submitted 2022-11-21; First posted 2022-12-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Bipolar Disorder Type II; Mood Depressive Disorder
Keywords: Bipolar disorder; Mood depressive disorder; RMN exploration; Metabolites concentration
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bipolar disorder group (Experimental): Patients with a diagnosis of bipolar II mood disorder stabilized in remission, according to DSM 5 criteria, with mood stabilizer treatment (lithium, anticonvulsant or antipsychotic) at an effective dose, with possible antidepressant treatment (SSRI, SNRI, tricyclics )
  Interventions: Diagnostic Test: NMR spectrometry
- Mood depressive disorder group (Experimental): Patients with a diagnosis of unipolar mood disorder stabilized in remission, according to DSM 5 criteria, with or without antidepressant treatment (SSRI, SNRI, tricyclics)
  Interventions: Diagnostic Test: NMR spectrometry
- Healthy volunteer (Experimental): People for whom no psychiatric diagnosis can be retained, according to DSM 5 criteria and naïve to psychotropic treatments
  Interventions: Diagnostic Test: NMR spectrometry

INTERVENTIONS:
Diagnostic Test: NMR spectrometry — The MRI protocol will be carried out at 3 Tesla (3T) on a Siemens NMR imaging system (Magnetom Vida, Siemens Healthcare, Erlangen, Germany), the emission of radiofrequency waves and the reception of the signal will be done using a resonator in quadrature head (64-channel phase-array antenna). The MRI protocol will take place in two phases:
  * Realization of a morphological sequence for the identification of the zone of interest.
  * Acquisition of a 1D NMR spectrum in the ventral striatum (right and left).
  * Acquisition of a 1D NMR spectrum in the anterior cingulate cortex (right and left).
  * Acquisition of a 1D NMR spectrum in the prefrontal cortex (right and left).

SUMMARY:
The presented project is an open and controlled single-center prospective exploratory study, evaluating the metabolic concentrations in the ventral striatum (VS), the Anterior cingulate cortex (ACC) and the prefrontal cortex (PFC) on the left and on the right of patients in remission of unipolar mood disorder and type II bipolar mood disorder compared to each other and to healthy subjects using NMR spectrometric measurements. We hypothesize that there is a significant difference between the mean glutamate concentrations in the ventral striatum (right and left) of the two groups of unipolar and bipolar type II patients. The average glutamate concentration would be higher for participants in the group of type II bipolar patients.

DETAILED DESCRIPTION:
Depression meets the same clinical diagnostic criteria whether it is the expression of a bipolar or unipolar mood disorder. It is essential to distinguish between these two disorders because the pharmacological management of this episode and the follow-up of the patient will be different. The risk of iatrogenesis is significant if the diagnosis is incorrect. Currently, there is no biomarker that can help the clinician in his diagnostic approach and to differentiate between bipolar and unipolar mood disorder (Grande et al., 2016; Vieta et al., 2018).

Many research, particularly in neuroimaging, explore these mood disorders to identify morphological, functional and metabolic signatures both in the state phase and in the asymptomatic phase.

Functional imaging work, carried out at the Cardiff University Brain Research Imaging Center in Wales in collaboration with the team 7280 from Clermont Auvergne University, is part of this research. The object of this work was to study the dopaminergic system, and in particular the meso-cortico-limbic pathway, which is the anatomical and functional substrate of the reward circuit. The activity of this system, when measured on functional MRI in the ventral striatum during an activation paradigm of the "anticipation of a reward during a monetary task" type, shows variations in the disorders of mood, in the state phase as well as in the asymptomatic phase. These activation differences are significantly different between healthy, unipolar and bipolar asymptomatic subjects.

The cerebral neurochemical processes involved in the physiopathology of mood disorders being still little studied at the present time and in order to complete these observations, the measurement and comparison of the concentrations of metabolites by NMR spectroscopy in these same regions (the meso -cortico-limbic) and under these same conditions will make it possible to specify the physiopathology of mood disorders. NMR spectroscopy, unlike functional MRI, allows us not only to compare groups, but also to measure concentrations in absolute values. Data from the literature show that these explorations are feasible in humans and meta-analyses suggest that a direct comparison could make it possible to discriminate mood disorders by the clinical dimension "capacity to experience pleasure" - or "hedonic capacity".

We hypothesize that there is a significant difference between the mean glutamate concentrations in the ventral striatum (right and left) of the two groups of unipolar and bipolar type II patients. The average glutamate concentration would be higher for participants in the group of type II bipolar patients.

This exploratory study will allow a better understanding of the pathophysiological mechanisms involved in the development of mood disorders and in particular in their clinical dimension "hedonic capacity", as well as to test the relevance of this potential biomarker (glutamate) than the current state of Art allows us to consider. The measurements in the control group will allow us to approach the values of the physiological norm. The measurements in the clinical groups will allow us to understand whether the "mood disorder" condition, even in remission, constitutes a sufficient factor of variation in this standard to allow them to be detected. This work would represent a first fundamental step in the understanding of pathophysiological mechanisms and the establishment of this measure as a biomarker for screening mood disorders and for discriminating between a unipolar disorder and a bipolar disorder and could thus guide the clinician in his diagnostic and therapeutic approach.

The constraints for the participants will be minimal with only two visits to the CHU. A first for the inclusion of a duration of 60 minutes. A second for the 120-minute measurement visit. The inclusion of patients will be done if possible during their regular follow-up to limit travel. Since MRI is a non-invasive technique used routinely in hospital practice, the risks incurred by patients are almost nil, subject to compliance with the contraindications of MRI

ELIGIBILITY:
BIPOLAR DISORDERS GROUP :

Inclusion criteria :

* Patients with a diagnosis of bipolar type II disorder stabilized in remission, according to DSM 5 criteria, with mood stabilizer treatment (lithium, anticonvulsant or antipsychotic) at an effective dose, with possible antidepressant treatment (SSRI, SNRI, tricyclics )
* Right handed
* Aged 18 to 40
* Having completed the MRI compatibility questionnaire and having no contraindication to MRI
* Having given their written, free and informed consent
* Affiliated to a social security scheme
* Effective contraception for participants of childbearing age
* ECOG performance index < 2

Exclusion criteria :

* Age < 18 or > 40
* BMI > 30kg/m2
* Current episode. (MADRS score > 15 or YMRS score > 12, Montgomery, 1979, Young et al, 1978)
* Unbalanced psychiatric pathology.
* Neurological pathology (e.g. parkinsonian syndrome, stroke, migraine, fibromyalgia, etc.)
* Psychiatric pathology other than bipolar mood disorder (e.g. schizophrenia, severe anxiety disorder, severe personality disorder, instinctual behavior disorder, autism spectrum disorder, disorder related to the use of psychoactive substances excluding tobacco.)
* Under current psychotropic treatment other than antidepressants (SSRI, SNRI, tricyclics) or mood stabilizer (lithium, anticonvulsant or antipsychotic) at an effective dose. Treatment with benzodiazepine possible if possibility of deferring this line of treatment when carrying out the NMR acquisition.
* Alcohol consumption >3 units of alcohol/day (30g/day) for men and >2 units of alcohol/day (20g/day) for women.
* Unbalanced progressive condition (hepatic failure, renal failure with creatinine clearance <30mL/min, respiratory failure, congestive heart failure, myocardial infarction during the last 6 months, etc.)
* Any active cancer
* Holders of a pacemaker, cochlear implants, metallic implants or any magnetic element
* Claustrophobia
* Pregnant and breastfeeding women
* Legal incapacity (person deprived of liberty or under guardianship)
* Who, for psychological, social, family or geographical reasons, cannot be followed and/or compliant with the requirements of the study
* Already included in another clinical trial

MOOD DEPRESSIVE DISORDERS GROUP :

Inclusion criteria :

* Patients with a diagnosis of unipolar mood disorder stabilized in remission, according to DSM 5 criteria, with or without antidepressant treatment (SSRI, SNRI, tricyclics)
* Right handed
* Aged 18 to 40
* Having completed the MRI compatibility questionnaire and having no contraindication to MRI
* Having given their written, free and informed consent
* Affiliated to a social security scheme
* Effective contraception for participants of childbearing age
* ECOG performance index < 2

Exclusion criteria :

* Age < 18 or > 40
* BMI > 30kg/m2
* Current episode. (MADRS score > 15 or YMRS score > 12, Montgomery, 1979, Young et al, 1978)
* Unbalanced psychiatric pathology.
* Neurological pathology (e.g. parkinsonian syndrome, stroke, migraine, fibromyalgia, etc.)
* Psychiatric pathology other than mood depressive disorder (e.g. schizophrenia, severe anxiety disorder, severe personality disorder, instinctual behavior disorder, autism spectrum disorder, disorder related to the use of psychoactive substances excluding tobacco.)
* Under current psychotropic treatment other than antidepressants (SSRI, SNRI, tricyclics) or mood stabilizer (lithium, anticonvulsant or antipsychotic) at an effective dose. Treatment with benzodiazepine possible if possibility of deferring this line of treatment when carrying out the NMR acquisition.
* Alcohol consumption >3 units of alcohol/day (30g/day) for men and >2 units of alcohol/day (20g/day) for women.
* Unbalanced progressive condition (hepatic failure, renal failure with creatinine clearance <30mL/min, respiratory failure, congestive heart failure, myocardial infarction during the last 6 months, etc.)
* Any active cancer
* Holders of a pacemaker, cochlear implants, metallic implants or any magnetic element
* Claustrophobia
* Pregnant and breastfeeding women
* Legal incapacity (person deprived of liberty or under guardianship)
* Who, for psychological, social, family or geographical reasons, cannot be followed and/or compliant with the requirements of the study
* Already included in another clinical trial

HEALTHY GROUP :

Inclusion criteria :

* People for whom no psychiatric diagnosis can be retained, according to DSM 5 criteria, naïve to psychotropic treatments
* Right handed
* Aged 18 to 40
* Having completed the MRI compatibility questionnaire and having no contraindication to MRI
* Having given their written, free and informed consent
* Affiliated to a social security scheme
* Effective contraception for participants of childbearing age
* ECOG performance index < 2

Exclusion criteria :

* Age < 18 or > 40
* BMI > 30kg/m2
* Current episode. (MADRS score > 15 or YMRS score > 12, Montgomery, 1979, Young et al, 1978)
* Unbalanced psychiatric pathology.
* Neurological pathology (e.g. parkinsonian syndrome, stroke, migraine, fibromyalgia, etc.)
* Psychiatric pathology (e.g. bipolar disorder, mood depressive disorder, schizophrenia, severe anxiety disorder, severe personality disorder, instinctual behavior disorder, autism spectrum disorder, disorder related to the use of psychoactive substances excluding tobacco.)
* Under current psychotropic treatment other than antidepressants (SSRI, SNRI, tricyclics) or mood stabilizer (lithium, anticonvulsant or antipsychotic) at an effective dose. Treatment with benzodiazepine possible if possibility of deferring this line of treatment when carrying out the NMR acquisition.
* Alcohol consumption >3 units of alcohol/day (30g/day) for men and >2 units of alcohol/day (20g/day) for women.
* Unbalanced progressive condition (hepatic failure, renal failure with creatinine clearance <30mL/min, respiratory failure, congestive heart failure, myocardial infarction during the last 6 months, etc.)
* Any active cancer
* Holders of a pacemaker, cochlear implants, metallic implants or any magnetic element
* Claustrophobia
* Pregnant and breastfeeding women
* Legal incapacity (person deprived of liberty or under guardianship)
* Who, for psychological, social, family or geographical reasons, cannot be followed and/or compliant with the requirements of the study
* Already included in another clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Glutamate concentration in ventral striatum | Within 3 months after inclusion
  The main objective of the study is to compare the mean concentrations of glutamate in the ventral striatum (right and left), between two groups of treated, asymptomatic patients: unipolar vs bipolar type II disorder. Patients will also be compared to a sample of healthy controls.

SECONDARY OUTCOMES:
Metabolites concentration in interest structures | Within 3 months after inclusion
  Comparison of mean concentrations of metabolites (Choline, myo-inositol, N-acetylaspartate, creatine, glutamate/glutamine, lactate, taurine, GABA) in the Ventral Striatum (VS), Anterior Cingulate Cortex (ACC) and Prefrontal Cortex (PFC) ) between the three groups
Metabolites relationships with Seniority, severity of the disorder | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Seniority, severity of the disorder measured by MADRS questionnaire
Metabolites relationships with Predominant polarity | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Predominant polarity by YMRS questionnaire
Metabolites relationships with Dimension Anhedonia | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Dimension Anhedonia by SHAP questionnaire
Metabolites relationships with Operation | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Operation by FAST questionnaire
Metabolites relationships with Quality of life by MARS questionnaire | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Quality of life
Metabolites relationships with Compliance with treatment | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Compliance with treatment by WHOQOL-BREF questionnaire
Metabolites relationships with description ofPharmacological class of the antidepressant | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with Pharmacological class of the antidepressant by
Metabolites relationships with description of Pharmacological class of mood stabilizer. | Within 3 months after inclusion
  Study of the relationships between the concentrations of metabolites with description of Pharmacological class of mood stabilizer.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne ALLAUZE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France